CLINICAL TRIAL: NCT06976294
Title: The Effect of Cognitive Behavioral Approach-Based Psychoeducation on Post-Traumatic Growth, Psychological Resilience, and Ruminative Thoughts in Primary Caregivers of Individuals Diagnosed With Alzheimer's Disease
Brief Title: The Effects of Cognitive Behavioral Approach-Based Psychoeducation on Caregivers of Alzheimer's Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Pınar Sevda Bozkurt, PhD student, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PAU-SBF-PSB-01
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Disease, Posttraumatic Growth
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary Caregivers of Individuals Diagnosed with Alzheimer's (Experimental group) (Experimental)
  Interventions: Other: Cognitive Behavioral Approach-Based Psychoeducation
- Primary Caregivers of Individuals Diagnosed with Alzheimer's (Control group) (No Intervention)

INTERVENTIONS:
Other: Cognitive Behavioral Approach-Based Psychoeducation — The 'Socio-Demographic Characteristics Form', the 'Post-Traumatic Growth Inventory', the 'Psychological Resilience Scale for Adults', and the 'Event-Related Rumination Inventory' will be administered to individuals in both the intervention and control groups. No intervention will be applied to the control group. For the intervention group, psychoeducation groups based on the cognitive behavioral approach will be formed for the primary caregivers. Eight face-to-face sessions, each lasting 60 to 90 minutes, will be conducted
  Arms: Primary Caregivers of Individuals Diagnosed with Alzheimer's (Experimental group)

SUMMARY:
Alzheimer's disease is a progressive and chronic neurocognitive disorder. Individuals who assume the role of primary caregivers and are responsible for meeting the care needs of the patient often develop serious health problems over time. It is particularly important to assess the psychological resilience of those who struggle to manage the caregiving process, to identify ruminative thoughts developed in response to negative experiences, and ultimately to determine the presence of post-traumatic growth. Cognitive Behavioral Therapy (CBT)-based psychoeducational interventions are highly effective in the holistic assessment and support of primary caregivers.

DETAILED DESCRIPTION:
Alzheimer's disease is a progressive and chronic neurocognitive disorder characterized by the deterioration of higher-level cortical functions, leading to cognitive decline, neuropsychiatric behavioral changes, and a reduced ability to perform daily activities. As the disease progresses, patients gradually lose functional abilities, resulting in an increased demand for care. Primary caregivers, who are directly responsible for meeting these care needs, often face significant emotional, physical, social, and financial burdens. Providing long-term care to elderly individuals is a major source of chronic stress and can exceed caregivers' coping capacities. In this context, psychological resilience serves as a critical protective factor. Interventions that enhance the resilience of caregivers supporting individuals with chronic mental illness are essential for caregiver empowerment. Caregivers with low resilience are more prone to maladaptive coping mechanisms, such as ruminative thinking. Rumination can intensify psychological distress when negative thoughts interact with depressive mood states during the processing of traumatic experiences. However, not all traumatic experiences lead to negative outcomes; in some cases, individuals may grow stronger and experience positive psychological changes, known as post-traumatic growth (PTG). PTG refers to the positive transformation that can emerge from the struggle with highly challenging life circumstances. The psychological toll of caregiving highlights the importance of supportive psychological interventions. Psychoeducational programs based on Cognitive Behavioral Therapy (CBT) offer a comprehensive approach by addressing the needs of caregivers while also considering both the patients and the broader family systems. This study aims to examine the effects of CBT-based psychoeducation on post-traumatic growth, psychological resilience, and ruminative thinking among primary caregivers of individuals diagnosed with Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Willing to participate in the study
* A member of the Denizli Alzheimer Association
* At least a primary school graduate
* Able to communicate effectively
* Providing primary care to an individual diagnosed with Alzheimer's for at least one year
* Providing primary care to a patient diagnosed with moderate to advanced stage Alzheimer's
* Serving as a primary caregiver for at least six months

Exclusion Criteria:

* Primary caregivers who have participated in any psychoeducation group
* Caregivers who have been diagnosed with any mental health disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Socio-Demographic Characteristics Form | two weeks
  It consists of questions covering descriptive characteristics of the primary caregivers of Alzheimer's patients, such as age, gender, education level, degree of relationship with the patient, and the duration of caregiving.

SECONDARY OUTCOMES:
Post-Traumatic Growth Inventory | two weeks
  The inventory consists of 21 items and five factors. It is a self-report scale in a five-point Likert format, scored between '0 (I did not experience this change)' and '5 (I experienced this change to a very great degree)'. The total score that can be obtained from the inventory ranges from 0 to 105. Higher scores indicate greater post-traumatic growth
Psychological Resilience Scale for Adults | two weeks
  The scale consists of a total of 33 items. Each item presents two opposing statements regarding a specific situation, and respondents are asked to mark the option that best reflects their level of agreement or appropriateness.
Event-Related Rumination Inventory | two weeks
  The inventory consists of 20 items and is divided into two sections of 10 items each, assessing two types of rumination: 'intrusive' and 'deliberate'. It is structured as a 4-point Likert scale, where a score of 0 indicates 'never' and a score of 3 indicates 'often.
Beck Depression Inventory | two weeks
  It is a 21-item assessment scale that measures depressive symptoms and characteristic attitudes. It uses a 4-point Likert-type format, with each item scored between 0 and 3. The total score ranges from 0 to 63.
Beck Anxiety Inventory | two weeks
  It is a 21-item assessment scale. Each item includes four options scored from 0 to 3. The total score from the 21 items ranges from 0 to 63, with higher scores indicating increased anxiety symptoms.